CLINICAL TRIAL: NCT03238378
Title: SALVAGE BRACHYTHERAPY WITH INTERSTITIAL HYPERTHERMIA FOR LOCALLY RECURRENT HEAD & NECK CARCINOMA FOLLOWING PREVIOUSLY EXTERNAL BEAM RADIATION THERAPY: A PROSPECTIVE PHASE II STUDY
Brief Title: Salvage Brachytherapy and Hyperthermia for Recurrent H&N-tumours
Acronym: HyBT-H&N
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Vratislav Strnad, Head of the Interstitial Brachytherapy at the Dept. of Radiooncology, University of Erlangen-Nürnberg Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HyBT-H&N
Record Dates: First submitted 2017-07-31; First posted 2017-08-03 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Locally Recurrent Head and Neck Cancer
Keywords: head and neck cancer; Locally recurrent head and neck cancer; Brachytherapy; Hyperthermia
MeSH Terms: conditions — Head and Neck Neoplasms; Hyperthermia | interventions — Brachytherapy; Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapy (Experimental): Brachytherapy d1-5(6) Hyperthermia d2 + 5
  Interventions: Radiation: Brachytherapy; Other: Hyperthermia

INTERVENTIONS:
Radiation: Brachytherapy — Brachytherapy d 1-5(6)
Other: Hyperthermia — Hyperthermia d 2 + 5

SUMMARY:
The aim of the present trial is to assess the prospective results of protocol-based interstitial pulsed-dose-rate (PDR) brachytherapy with interstitial hyperthermia (iHT) in a group of selected patients where salvage surgery with clear resection margins was not possible.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent carcinoma of the head and neck region
* Stage rcT1-3
* Tumor anatomy and location suitable for brachytherapy techniques.
* cN0/pN0 or rpN+ & R0 with <3 pos. LND & without invasion of capsula.
* M0
* ECOG 0-2
* Previous radiation therapy up to at least 50 Gy
* Previous radiation therapy completed more than 6 months ago
* Written study-specific informed consent

Exclusion Criteria:

* cT4
* rpN+ with >2 pos. LND or invasion of capsula
* Pregnant or lactating women
* Collagen vascular disease
* The presence of congenital diseases with increased radiation sensitivity, for example Ataxia telangiectatica or similar
* Psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2017-03-29 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Late side effects | Effects are followed up to 5 years after therapy
  Comparison late side effects to standard therapy

SECONDARY OUTCOMES:
Quality of life | up to 5 years after therapy
  Assessment of quality of life with EORTC questionnaires
Rate of local recurrencies | up to 5 years after therapy
  Assessment of cumulative local recurrence rate
Overall survival | up to 5 years after therapy
  Rate of Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Vratislav Strnad, MD, Principal Investigator — Dept. of Radiation Therapy, University Hospital Erlangen
Locations (1):
- Dept. of Radiation Therapy, University Hospital Erlangen, Erlangen, Germany